CLINICAL TRIAL: NCT04886297
Title: Department of Nutrition and Food Hygiene,School of Public Health, Sun Yat-sen University
Brief Title: A Dose-response Study of Dietary Resveratrol on Lipid Metabolism Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Yuqing, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: lwh87331597
Record Dates: First submitted 2021-05-07; First posted 2021-05-14 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- placebo (Placebo Comparator): The placebo capsules only contained pullulan and maltodextrin. During the trial period, the participants were instructed to consume two Mega Resveratrol® placebo capsules once daily (30 min after breakfast).
  Intervention: Drug: Mega Resveratrol® capsules
  Interventions: Drug: Mega Resveratrol® Placebo capsules
- 100mg/d resveratrol (Experimental): During the trial period, the participants will be instructed to consume one Mega Resveratrol® capsules and one Mega Resveratrol® placebo capsules 30 min after breakfast. The resveratrol capsules (100 mg anthocyanins per capsule) will provid a total daily intake of 100 mg resveratrol.
  Intervention: Drug: Mega Resveratrol® capsules
  Interventions: Drug: Mega Resveratrol® capsules
- 300mg/d resveratrol (Experimental): During the trial period, the participants will be instructed to consume one Mega Resveratrol® capsules and one Mega Resveratrol® placebo capsules 30 min after breakfast. The resveratrol capsules (300 mg anthocyanins per capsule) will provid a total daily intake of 300 mg resveratrol.
  Intervention: Drug: Mega Resveratrol® capsules
  Interventions: Drug: Mega Resveratrol® capsules
- 600mg/d resveratrol (Experimental): During the trial period, the participants will be instructed to consume two Mega Resveratrol® capsules 30 min after breakfast. The resveratrol capsules (300 mg anthocyanins per capsule, 2 per day) will provid a total daily intake of 600 mg resveratrol.
  Intervention: Drug: Mega Resveratrol® capsules
  Interventions: Drug: Mega Resveratrol® capsules

INTERVENTIONS:
Drug: Mega Resveratrol® capsules — Subjects were orally administered Mega Resveratrol® capsules daily for 8 weeks.
  Arms: 100mg/d resveratrol; 300mg/d resveratrol; 600mg/d resveratrol
Drug: Mega Resveratrol® Placebo capsules — Mega Resveratrol® Placebo capsules
  Arms: placebo

SUMMARY:
In order to study the effect of resveratrol on the improvement of lipid and uric acid metabolism, randomized intervention trials were conducted to compare the effects of resveratrol on the improvement of lipid and uric acid metabolism in different dose groups. To explore the best dose of resveratrol for the prevention and treatment of metabolic diseases provide an important scientific basis.

DETAILED DESCRIPTION:
In order to study the effect of resveratrol on the improvement of lipid and uric acid metabolism, randomized controlled trials were conducted to enrolled 160 patients with dyslipidemia. The subjects were divided into 0 mg / d, 100 mg / d, 300 mg / d, 600 mg/ d four dose groups, intervention for 8 weeks, comparing different doses of resveratrol on lipid and uric acid metabolism. To explore the best dose of resveratrol for the prevention and treatment of metabolic diseases provide an important scientific basis.

ELIGIBILITY:
Inclusion Criteria:

* Dyslipidemia
* The age between 35 and 70 years old

Exclusion Criteria:

* Intake of any medicine that affect lipid metabolism currently or in the preceding 6 months
* Dietary supplementation with phytochemicals including resveratrol in the preceding 3 months
* History of acute or chronic infectious disease, autoimmune disease, cancer, traumatic injury, or surgery in the preceding 1 month
* History of severe chronic disease including AS and CVD, liver or renal dysfunction, and lactation or pregnancy
* Pregnant woman and Breast Feeding Women

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Effect of resveratrol on lipid profile in patients with dyslipidemia | Change from Baseline to 4 weeks and 8 weeks
  Lipid profile in serum will be measured, mainly including TC, TG, LDL-C and HDL-C, by automatic biochemical analyzer.

SECONDARY OUTCOMES:
Effect of resveratrol on uric acid and xanthine oxidase in patients with dyslipidemia | Change from Baseline to 4 weeks and 8 weeks
  Uric acid concentration and xanthine oxidase activity will be measured by automatic biochemical analyzer and commercial kits, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Wenhua, Principal Investigator — North Campus, Guangzhou Campus, No. 74, Zhongshan 2nd Road, Yuexiu District, Guangzhou
Locations (1):
- Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou Y, Zeng Y, Pan Z, Jin Y, Li Q, Pang J, Wang X, Chen Y, Yang Y, Ling W. A Randomized Trial on Resveratrol Supplement Affecting Lipid Profile and Other Metabolic Markers in Subjects with Dyslipidemia. Nutrients. 2023 Jan 17;15(3):492. doi: 10.3390/nu15030492. PMID 36771199